CLINICAL TRIAL: NCT02326376
Title: Non-interventional PASS to Evaluate Safety of Kineret in Treatment of CAPS in Routine Clinical Care With Regard to Serious Infections, Malignancies, Injection Site Reactions, Allergic Reactions, Medication Errors Including Re-use of Syringe
Brief Title: Kineret CAPS Post Authorisation Study
Status: Completed | Type: Observational
Sponsor: Swedish Orphan Biovitrum (Industry)
Collaborators: Pediatric Rheumatology International Trials Organization (Other)
Responsible Party: Sponsor
Other Study IDs: Sobi.Anakin-201; ENCEPP/SDPP/6366 (Registry Identifier: EU PAS Registry No)
Record Dates: First submitted 2014-12-01; First posted 2014-12-29 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Cryopyrin-Associated Periodic Syndromes
MeSH Terms: conditions — Cryopyrin-Associated Periodic Syndromes | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CAPS patients: CAPS patients treated with anakinra, using the Kineret graduated syringe
  Interventions: Drug: anakinra (Kineret)

INTERVENTIONS:
Drug: anakinra (Kineret)
  Other Names: Kineret

SUMMARY:
A non-interventional, post authorization safety study to evaluate the safety of Kineret in the treatment of Cryopyrin Associated Periodic Syndromes (CAPS) in routine clinical care with regard to serious infections, malignancies, injection site reactions, allergic reactions and medication errors, including re-use of syringe.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent by the patient and/or caregiver
* Kineret treatment will be according to the Summary of Product Characteristics (SmPC), as confirmed by the Investigator

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All CAPS patients treated with Kineret at the selected sites.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2015-04-24 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2019-09-12 (Actual)

PRIMARY OUTCOMES:
Rate of serious infections | 3 years
Rate of new malignancies | 3 years
Rate of injection site reactions | 3 years
Rate of allergic reactions | 3 years
Rate of medication errors including re-use of syringe | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Marco Gattorno, MD, Principal Investigator — IRCCS Istituto Giannina Gaslini; Torbjörn Kullenberg, MD, Study Director — Swedish Orphan Biovitrum AB (publ)
Locations (2):
- Swedish Orphan Biovitrum Investigational Site, Groningen, Netherlands
- Swedish Orphan Biovitrum Investigational Site, London, United Kingdom